CLINICAL TRIAL: NCT06408441
Title: The Observational EURACAN Prospective Clinical Registry Dedicated to Epithelioid Hemangioendothelioma: the Protocol of an International and Collaborative Effort on an Ultra-rare Entity
Brief Title: The Epithelioid Hemangioendothelioma Registry of the European Reference Network on Rare Adult Solid Cancers (EURACAN)
Acronym: EHE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Annalisa Trama, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT 43-21
Record Dates: First submitted 2024-04-03; First posted 2024-05-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Epithelioid Hemangioendothelioma; Sarcoma,Soft Tissue
Keywords: rare cancers; soft tissue rare cancer; registry; protocol; ultra rare sarcomas
MeSH Terms: conditions — Hemangioendothelioma, Epithelioid; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — Tumour and healthy biological samples (paraffin-embedded or fresh tissue, blood) previously collected in the course of routine health care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- unifocal disease: Primary, localized, single lesion
- Loco-regional disease: multifocal single-organ involvement
- Systemic metastases: multi-organ involvement and/or loco-regional lymph-node involvement

SUMMARY:
Epithelioid hemangioendothelioma (EHE) is an ultra-rare sarcoma, marked by distinctive molecular and pathological features and with a variable clinical behavior. Its natural history is still partially understood, reliable prognostic and predictive factors are lacking and many questions are still open on the optimal management. In the context of EURACAN, a prospective registry specifically dedicated to EHE was developed and launched with the aim of providing, through high-quality prospective data collection, a better understanding of this disease.

The study design is a registry-based cohort study including only new cases of patients with a pathological and molecularly confirmed diagnosis of EHE.

The objectives are to improve the understanding of EHE natural history, validate and identify new prognostic and predictive factors, clarify the activity and efficacy of currently available treatment options, describe treatment pattern.

It is an hospital-based registry established in centres with expertise in EHE including adult patients with a new pathological and molecularly confirmed diagnosis of EHE starting from the 1st December 2023. The characteristics of each patient in the facility who meets the above-mentioned inclusion criteria will be collected prospectively and longitudinally with follow-up at cancer progression and / or cancer relapse or patient death.

The data analyses will include descriptive statistics and analytical analyses. Multivariable Cox's proportional hazards model and Hazard ratios (HR) for all-cause or cause-specific mortality will be used to determine independent predictors of overall survival, recurrence and progression.

The registry has been joined by 21 sarcoma reference centers across EU and UK, covering 10 countries. Patients' recruitment started in December 2023. The estimated completion date is December 2033 upon agreement on the achievement of all the registry objectives. The already established collaboration and participation of EHE patient's associations involved in the project will help in promoting the registry and fostering accrual.

This registry has been developed with the support of EHE Rare Cancer Charity UK, STATER (Grant Agreement number: 947604, HP-PJ-2019) and EURACAN 2022 (Grant Agreement number: 101085486, EU4H-2022-ERN-IBA) European Health and Digital Executive Agency (HaDEA)

DETAILED DESCRIPTION:
Given its incidence of 0.038/100 000/year, EHE is an ultra-rare sarcoma, with distinctive, well-defined pathological, molecular and clinical features. It belongs to the group of vascular sarcomas and is characterized by WWTR1-CAMTA1 (90%) or YAP1-TFE3 (10%) gene fusions, which represents today a hallmark for diagnosis. EHE potentially arises everywhere in the body and shows a high tendency toward metastatic spread, especially in the lung, liver and bone. The onset is characterized by different presentations, including a unifocal lesion (usually in the soft tissues), locoregional metastases (multiple lesions in a single organ or in a single anatomic compartment) and systemic metastases (multi-organ involvement). Also, the biological behavior of the disease is unique in sarcomas and variable, with spontaneous regressions reported, patients with untreated stable disease overtime, slowly progressive variants and highly aggressive and rapidly fatal cases. Today, the relative incidence of the different presentations is undefined, the natural history of the different subtypes is poorly understood, and reliable clinical or biological prognostic factors are lacking. Retrospective data suggest that patients with EHE presenting or developing during their course serosal involvement and / or effusion, systemic associated symptoms and anemia have a worse prognosis, but a prospective validation of this observation is lacking. In terms of management, surgery is the treatment of choice for localized disease, with an excellent outcome (expected cure rate of 70-80%) and no proven role for local or systemic adjuvant therapies. For patients with advanced, asymptomatic disease, active surveillance is often the upfront choice in order to minimize the risk of overtreatment. Systemic therapies are usually considered for patients with progressive or symptomatic disease, although a standard medical approach is currently not established. Unfortunately, conventional chemotherapy, including anthracycline-based regimens widely regarded as the mainstay in the treatment of advanced soft tissue sarcomas, showed marginal activity in EHE. The use of potentially active compounds, such as m-TOR inhibitors which proved the highest activity in EHE and could therefore represent the preferred option, is limited by regulatory constraints as they are not currently labeled in Europe for this indication. Given the degree of uncertainty on EHE management, a global consensus meeting was organized in December 2020 under the umbrella of the European Society for Medical Oncology (ESMO) involving > 80 multidisciplinary, worldwide experts together with a patient representative, with the aim of defining, by consensus, evidence-based best practices for the optimal approach to primary and metastatic EHE.

Since the number of patients is inherently low at the hospital level, the only way to increase knowledge about EHE and improve the diagnosis, treatment, and prognosis of this complex and heterogeneous disease is to harmonize and combine real-world data from sarcoma expert centres by leveraging a wide, international, joined effort. In this context, a unique opportunity is provided by the European Reference Networks (ERNs), virtual network established by the EU commission aiming to tackle rare conditions, including cancers. Among the three ERNs dedicated to cancer, EURACAN (https://euracan.eu) is the one focusing on the 10 families of rare adult solid cancers (RACs), including soft tissue sarcomas, bone sarcomas and gastrointestinal stromal tumour. Fostering academic research and promote epidemiological surveillance in rare cancers through setting up of shared registries is recognize as one of ERNs priorities. Within the sarcoma domain, taking into account the challenges described above, priority was given to ultra-rare sarcoma, and thanks to the strong connection, motivation and support provided by EHE Rare Cancer Charity UK, it was decided to start from EHE. We believe that in this context the collection of high-quality data by clinical registries will be crucial to improve the understanding of EHE natural history, validate and identify new prognostic factors, clarify the activity and efficacy of currently available treatment options and eventually provide and external control which might serve as a benchmark for the development of new drugs and support discussion with regulatory authorities.

The EURACAN EHE registry is a prospective clinical registry that will collect data from all new patients receiving a pathological and molecularly confirmed diagnosis of EHE starting from the 1st December 2023. To this aim, an EHE-focused clinical record form (CRF) was developed through the Research Electronic Data Capture (REDCap) and designed to capture the specific features of this disease.

For each patient, data collection will include:

1. A common baseline, including full details on demographic, comorbidities (special focus on immune-mediated and gynecological diseases), concomitant medications, physical examination, systemic symptoms at presentation, tumour-related pain assessment, blood tests, pathology and molecular features (on the diagnostic specimen), EHE extension at baseline (unifocal disease, loco-regional disease, systemic metastases)
2. Depending on the disease extent, detail on staging modalities, primary site and size, extension of metastatic disease (organs involved, number of lesions), presence and characterization of serosal involvement and effusion, treatment (surgery, radiation therapy, medical therapies, isolated limb perfusion, other locoregional techniques).

Although the EHE registry per se does not foresee any collection of pathological samples and / or imaging, the availability for each enrolled patient of pathological samples, massive parallel sequencing data and imaging at the contributing institution will be captured by the CRF, in order to facilitate patients' identification for future dedicated studies which will imply the use of these data.

Given the peculiar biological EHE behavior, in absence of any event, a mandatory 6-monthly update will be required at all contributing centers. In the mandatory 6-monthly update, information from the last visit will be recorded regarding: physical examination, time interval of development of systemic symptoms, assessment of tumor-related pain, blood tests, update on ongoing treatment / active surveillance (including modalities and timing of radiological monitoring and radiological response).

All events will be recorded at the time of the occurrence (for unifocal disease, local recurrence and metastatic progression; for locoregional and metastatic disease, systemic progression). For every event, information will be recorded on physical examination, time interval of development of systemic symptoms, assessment of tumor-related pain assessment, blood tests (hemoglobin and fibrinogen), radiological modalities detecting progression, extent of progression (by RECIST 1.1 and not), serosal involvement and / or effusion, update on ongoing treatment / active surveillance.

Patient status (alive with no evidence of disease, alive with disease, dead) and last follow up will be updated at any data entry.

The registry and therefore the electronic CRF have been shaped starting from what have been agreed and reported in the EHE consensus paper from the sarcoma community of experts, published in 2021. A registry kick-off meeting was held in Milan the 15th September 2023, involving the EHE prospective clinical registry coordination team, all the contributing centers and patients' associations (EHE Rare Cancer Charity UK, EHE Italia and EHE US) to present the registry and share common clinical practice guidelines, derived from the consensus paper, to be followed for the patients with EHE included in the registry.

The launch of the EHE prospective clinical registry was shared with all the reference institutions belonging as full members or associated partners to EURACAN sarcoma domain (63 institutions across Europe).

The project was also opened to EU institutions not belonging to EURACAN and extra-EU institutions. In this case, in order to ensure an adequate degree of expertise in the disease, the institutions interested in joining the registry were asked to provide the number of new EHE cases (molecularly confirmed) seen each year over 3 years (2020-2021-2022) and a threshold of at least 20% of EHE national incident cases was selected for participation.

As a result of this process, 21 institutions joined the registry in September 2023, 17 of which belonging to EURACAN, from 10 countries.

The registry is federated thus, data are stored by the health care providers contributing to the registry. At the local level, data are pseudonymised.

Statistical analyses will be performed based on a study protocol. Queries will be developed, in collaboration with clinical experts, to interrogate the EURACAN EHE registry to generate the descriptive statistics and relevant information needed to plan the analyses envisaged by the study protocol.

Data quality checks aim to assess whether data values are present, if they adhere to specific standard and if they are believable in terms of:

* Conformance: the data should be recorded in agreement with the correct formats (e.g. range of values, date formats);
* Completeness: the data should not have missing values or data records;
* Plausibility: the data should be believable (e.g. internal consistency; temporal and atemporal comparison);

Quality checks of the data conformance are included in the CRF in the form of predefined alerts and errors running during the data input. Moreover, several additional completeness and plausibility checks (e.g. completeness of variables for each patient, plausibility of temporal intervals between different dates, etc.) are implemented in an external web tool connected to the CRF by use of API key, capable of executing all data quality checks simultaneously. The API key is not transmitted outside the centre, it is used only locally to perform data quality checks. The results of these checks are available locally for each centre and periodically they will be summarized in reports that the registry coordination team (INT) will monitor and discuss with each centre.

Legal basis of the registry:

In Europe, the processing of personal data for scientific research can be grounded upon several conditions of lawfulness, established in Article 9(2) of the General Data Protection Regulation (GDPR). Among these, the most relevant ones are:

* the consent of data subjects (Art. 9(2)lit. a);
* the pursuing of a substantial public interest, on the basis of Union or Member State law (Art. 9(2)lit. g);
* the pursuing of a scientific research purpose on the basis of Union or Member State law (Art. 9(2)lit. j).

The GDPR allows or requires Member States to implement national specifications or derogations from certain rules set out in the GDPR, therefore the legal basis of the federated registry will be based in each participating hospital on the laws and regulations of its country.

ELIGIBILITY:
Inclusion Criteria:

* New patients managed by the contributing centers with a pathological EHE diagnosis performed or verified by an expert sarcoma pathologist starting from 1 December 2023 onwards and to be performed within 6 months from the registration
* Molecular confirmation of the diagnosis (WWTR1-CAMTA1 or YAP1-TFE3)
* Adult patients (aged ≥ 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is an hospital based registry thus, hospitals experts in rare cancer. This registry will not select a sample of patients, but it will include every accordant patient present in each facility.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2033-12-01 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Male to Female (M/F) ratio | 2 years
  Difference between the number of males and females
Age average | 2 years
  The mathematical average age of all the members of a population (i.e. EHE patients)
Comorbidity | 2 years
  Proportion of patients with Charlson Comorbidity Index (CCI) score mild (CCI scores of 1-2); moderate (CCI scores of 3-4); and severe (CCI scores ≥5)
Performance status | 2 years
  Proportion of patients by ECOG performance status grade
Cumulative incidence of local recurrence | 5 years
  proportion of cancer patients who develop a local recurrence over time
Cumulative incidence of distant metastasis | 5 years
  proportion of cancer patients who develop distant metastases over time
Time to local progression | 5 years
  Time elapsed from diagnosis to local progression
Time to distant metastases | 5 years
  Time elapsed from diagnosis to distant metastasis
Overall survival | 5 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive
Progression free survival | 5 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse
Treatment effectiveness | 2 years
  Competitive cumulative incidence of local recurrence and distant metastases
Disease free survival | 5 years
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
Description of treatment pattern and quality of care | 2 years
  Percentage of patients treated according to Consensus paper recommendations

CONTACTS AND LOCATIONS:
Locations (21):
- University Hospital Graz, Graz, Graz, Austria
- Aarhus University Hospital, Aarhus, Aarhus, Denmark
- Léon Bérard Center, Lyon, Lyon, France
- Essen University Hospital, Essen, Hesse, Germany
- Italy (10):
  - Istituto Ortopedico Rizzoli, Bologna, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Careggi, Firenze
  - IRCCS Istituto Clinica Humanitas, Rozzano, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan
  - Istituto Oncologico Veneto, Padua, Padova
  - Policlinico Universitario P. Giaccone, Palermo, Palermo
  - Nuovo Ospedale di Prato "S.Stefano", Prato, Prato
  - Università Campus Bio-Medico, Roma, Roma
  - Istituto Nazionale dei Tumori Regina Elena, Roma, Roma
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Torino
- Oslo University hospital Ullevål, Oslo, Oslo County, Norway
- Maria Skłodowska-Curie Institute of Oncology, Warsaw, Warsaw, Poland
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Göteborg
  - Karolinska University Hospital, Stockholm, Stockholm County
- The Royal Marsden Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The governance (link https://euracan.eu/registries/euracan-registry/registry-governance/) set the data access rules to the federated registry
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 5 years
Access Criteria: 1. data remain the contributing Health Care Providers (HCP)
  2. each HCP is free to access and use its own data for research
  3. each contributing HCP and third parties can request access to the database following the rules including in the governance

REFERENCES:
- [Background] Stacchiotti S, Frezza AM, Blay JY, Baldini EH, Bonvalot S, Bovee JVMG, Callegaro D, Casali PG, Chiang RC, Demetri GD, Demicco EG, Desai J, Eriksson M, Gelderblom H, George S, Gounder MM, Gronchi A, Gupta A, Haas RL, Hayes-Jardon A, Hohenberger P, Jones KB, Jones RL, Kasper B, Kawai A, Kirsch DG, Kleinerman ES, Le Cesne A, Lim J, Chirlaque Lopez MD, Maestro R, Marcos-Gragera R, Martin Broto J, Matsuda T, Mir O, Patel SR, Raut CP, Razak ARA, Reed DR, Rutkowski P, Sanfilippo RG, Sbaraglia M, Schaefer IM, Strauss DC, Sundby Hall K, Tap WD, Thomas DM, van der Graaf WTA, van Houdt WJ, Visser O, von Mehren M, Wagner AJ, Wilky BA, Won YJ, Fletcher CDM, Dei Tos AP, Trama A. Ultra-rare sarcomas: A consensus paper from the Connective Tissue Oncology Society community of experts on the incidence threshold and the list of entities. Cancer. 2021 Aug 15;127(16):2934-2942. doi: 10.1002/cncr.33618. Epub 2021 Apr 28. PMID 33910263
- [Background] Blay JY, Piperno-Neumann S, Watson S, Dufresne A, Valentin T, Duffaud F, Toulmonde M, Italiano A, Bertucci F, Tlemsani C, Firmin N, Bompas E, Perrin C, Ropars M, Saada-Bouzid E, Dubray-Longeras P, Hervieu A, Lebbe C, Gantzer J, Chaigneau L, Fiorenza F, Rios M, Isambert N, Soibinet P, Boudou-Roquette P, Verret B, Ferron G, Ryckewaert T, Lebellec L, Brahmi M, Gouin F, Meeus P, Vaz G, Le Loarer F, Karanian M, De Pinieux G, Ducimetiere F, Chemin C, Morelle M, Le Cesne A, Penel N; NETSARC/REPPS/RESOS and French Sarcoma Group-Groupe d'Etude des Tumeurs Osseuses (GSF-GETO) networks. Epithelioid hemangio-endothelioma (EHE) in NETSARC: The nationwide series of 267 patients over 12 years. Eur J Cancer. 2023 Oct;192:113262. doi: 10.1016/j.ejca.2023.113262. Epub 2023 Jul 29. PMID 37625241
- [Background] Stacchiotti S, Miah AB, Frezza AM, Messiou C, Morosi C, Caraceni A, Antonescu CR, Bajpai J, Baldini E, Bauer S, Biagini R, Bielack S, Blay JY, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brodowicz T, Callegaro D, De Alava E, Deoras-Sutliff M, Dufresne A, Eriksson M, Errani C, Fedenko A, Ferraresi V, Ferrari A, Fletcher CDM, Garcia Del Muro X, Gelderblom H, Gladdy RA, Gouin F, Grignani G, Gutkovich J, Haas R, Hindi N, Hohenberger P, Huang P, Joensuu H, Jones RL, Jungels C, Kasper B, Kawai A, Le Cesne A, Le Grange F, Leithner A, Leonard H, Lopez Pousa A, Martin Broto J, Merimsky O, Merriam P, Miceli R, Mir O, Molinari M, Montemurro M, Oldani G, Palmerini E, Pantaleo MA, Patel S, Piperno-Neumann S, Raut CP, Ravi V, Razak ARA, Reichardt P, Rubin BP, Rutkowski P, Safwat AA, Sangalli C, Sapisochin G, Sbaraglia M, Scheipl S, Schoffski P, Strauss D, Strauss SJ, Sundby Hall K, Tap WD, Trama A, Tweddle A, van der Graaf WTA, Van De Sande MAJ, Van Houdt W, van Oortmerssen G, Wagner AJ, Wartenberg M, Wood J, Zaffaroni N, Zimmermann C, Casali PG, Dei Tos AP, Gronchi A. Epithelioid hemangioendothelioma, an ultra-rare cancer: a consensus paper from the community of experts. ESMO Open. 2021 Jun;6(3):100170. doi: 10.1016/j.esmoop.2021.100170. Epub 2021 Jun 2. PMID 34090171
- [Background] Amin RM, Hiroshima K, Kokubo T, Nishikawa M, Narita M, Kuroki M, Nakatani Y. Risk factors and independent predictors of survival in patients with pulmonary epithelioid haemangioendothelioma. Review of the literature and a case report. Respirology. 2006 Nov;11(6):818-25. doi: 10.1111/j.1440-1843.2006.00923.x. PMID 17052315
- [Background] Stacchiotti S, Simeone N, Lo Vullo S, Baldi GG, Brunello A, Vincenzi B, Palassini E, Dagrada G, Collini P, Morosi C, Greco FG, Sbaraglia M, Dei Tos AP, Mariani L, Frezza AM, Casali PG. Activity of sirolimus in patients with progressive epithelioid hemangioendothelioma: A case-series analysis within the Italian Rare Cancer Network. Cancer. 2021 Feb 15;127(4):569-576. doi: 10.1002/cncr.33247. Epub 2020 Oct 27. PMID 33107985
- [Background] Frezza AM, Napolitano A, Miceli R, Badalamenti G, Brunello A, Buonomenna C, Casali PG, Caraceni A, Grignani G, Gronchi A, Infante G, Morosi C, Saita L, Simeone N, Zaffaroni N, Vincenzi B, Stacchiotti S. Clinical prognostic factors in advanced epithelioid haemangioendothelioma: a retrospective case series analysis within the Italian Rare Cancers Network. ESMO Open. 2021 Apr;6(2):100083. doi: 10.1016/j.esmoop.2021.100083. Epub 2021 Mar 10. PMID 33714008
- [Background] Frezza AM, Ravi V, Lo Vullo S, Vincenzi B, Tolomeo F, Chen TW, Teterycz P, Baldi GG, Italiano A, Penel N, Brunello A, Duffaud F, Hindi N, Iwata S, Smrke A, Fedenko A, Gelderblom H, Van Der Graaf W, Vozy A, Connolly E, Grassi M, Benjamin RS, Broto JM, Grignani G, Jones RL, Kawai A, Tysarowski A, Mariani L, Casali PG, Stacchiotti S. Systemic therapies in advanced epithelioid haemangioendothelioma: A retrospective international case series from the World Sarcoma Network and a review of literature. Cancer Med. 2021 Apr;10(8):2645-2659. doi: 10.1002/cam4.3807. Epub 2021 Mar 13. PMID 33713582
- [Background] Engel ER, Cournoyer E, Adams DM, Stapleton S. A Retrospective Review of the Use of Sirolimus for Pediatric Patients With Epithelioid Hemangioendothelioma. J Pediatr Hematol Oncol. 2020 Nov;42(8):e826-e829. doi: 10.1097/MPH.0000000000001643. PMID 31714437
- [Background] Shibayama T, Makise N, Motoi T, Mori T, Hiraoka N, Yonemori K, Watanabe SI, Esaki M, Morizane C, Okuma T, Kawai A, Ushiku T, Yatabe Y, Yoshida A. Clinicopathologic Characterization of Epithelioid Hemangioendothelioma in a Series of 62 Cases: A Proposal of Risk Stratification and Identification of a Synaptophysin-positive Aggressive Subset. Am J Surg Pathol. 2021 May 1;45(5):616-626. doi: 10.1097/PAS.0000000000001660. PMID 33729740
- [Background] Rosenbaum E, Jadeja B, Xu B, Zhang L, Agaram NP, Travis W, Singer S, Tap WD, Antonescu CR. Prognostic stratification of clinical and molecular epithelioid hemangioendothelioma subsets. Mod Pathol. 2020 Apr;33(4):591-602. doi: 10.1038/s41379-019-0368-8. Epub 2019 Sep 19. PMID 31537895
- [Background] Bagan P, Hassan M, Le Pimpec Barthes F, Peyrard S, Souilamas R, Danel C, Riquet M. Prognostic factors and surgical indications of pulmonary epithelioid hemangioendothelioma: a review of the literature. Ann Thorac Surg. 2006 Dec;82(6):2010-3. doi: 10.1016/j.athoracsur.2006.06.068. PMID 17126100
- [Background] Deyrup AT, Tighiouart M, Montag AG, Weiss SW. Epithelioid hemangioendothelioma of soft tissue: a proposal for risk stratification based on 49 cases. Am J Surg Pathol. 2008 Jun;32(6):924-7. doi: 10.1097/pas.0b013e31815bf8e6. PMID 18551749
- [Background] Antonescu CR, Le Loarer F, Mosquera JM, Sboner A, Zhang L, Chen CL, Chen HW, Pathan N, Krausz T, Dickson BC, Weinreb I, Rubin MA, Hameed M, Fletcher CD. Novel YAP1-TFE3 fusion defines a distinct subset of epithelioid hemangioendothelioma. Genes Chromosomes Cancer. 2013 Aug;52(8):775-84. doi: 10.1002/gcc.22073. Epub 2013 Jun 5. PMID 23737213
- [Background] Mentzel T, Beham A, Calonje E, Katenkamp D, Fletcher CD. Epithelioid hemangioendothelioma of skin and soft tissues: clinicopathologic and immunohistochemical study of 30 cases. Am J Surg Pathol. 1997 Apr;21(4):363-74. doi: 10.1097/00000478-199704000-00001. PMID 9130982